CLINICAL TRIAL: NCT00999167
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of HPN-100 for Maintaining Remission in Subjects With Cirrhosis and Episodic Hepatic Encephalopathy
Brief Title: A Study of Safety and Efficacy of HPN-100 in Subjects With Cirrhosis and Episodic Hepatic Encephalopathy
Acronym: HALT-HE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPN-100-008
Record Dates: First submitted 2009-10-08; First posted 2009-10-21 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
Keywords: Cirrhosis; Episodic Hepatic Encephalopathy; HE; HPN-100; GT4P; glycerol phenylbutyrate
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPN-100 (Experimental)
  Interventions: Drug: HPN-100
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPN-100 — Part B: 6 mL BID for 16 weeks.
  Other Names: GT4P
  Arms: HPN-100
Drug: Placebo — Part B: same as experimental arm
  Arms: Placebo

SUMMARY:
This is a phase 2 study of HPN-100 in subjects with hepatic encephalopathy (HE) consisting of an open label safety lead-in (Part A), followed by randomized, double-blind, placebo-controlled treatment (Part B).

DETAILED DESCRIPTION:
Part A: Open-label, dose-escalation lead-in to assess HPN-100 safety and PK Approximately 10 subjects with HE and cirrhosis classified as Child Pugh B or C will undergo a one-step dose escalation over 4 weeks. Subjects will initially receive 6 mL HPN-100 BID for 1 week. On Day 7 and following satisfactory safety assessment of the subject, the dose will be escalated to 9 mL BID for an additional 3 weeks.

In addition to a safety assessment, subjects will undergo 12-hour PK assessments on Days 7 and 28, with sampling at the following time points (relative to the first dose): 0 (pre-first daily dose of HPN-100), 2, 4, 8 (approximately 2 hours before the second daily dose of HPN 100), and 12 hours post-first dose (approximately 2 hours after the second daily dose of HPN-100). Additional PK samples will be collected on Days 8, 15, and 21 (at pre-first dose and 4 hours post-first dose).

The DSMB will review all safety information, including laboratory values, to determine if Part B may be initiated.

Subjects enrolled in Part A may be eligible for Part B as long as they meet the eligibility criteria.

Part B: Randomized, double-blind assessment of HPN-100 in HE subjects Subjects who meet all entry criteria and are judged to be compliant with their prescribed SOC will be eligible for randomization to receive either HPN-100 or matching placebo for 16 weeks. Efficacy will be assessed by the proportion of subjects experiencing episodes of HE, as well as by other outcome measures, including daily home assessments.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and over
* Clinical diagnosis of cirrhosis of any cause
* Potential to benefit from HE treatment
* History of greater than or equal to 2 documented episodes of WH Grade 2 or more HE within the past 6 months, at least one of which occurred within the preceding 3 months
* No change in other HE-specific medications within 1 week before randomization
* Able to give informed consent and comply with study activities
* Availability of at least one designated family member or caregiver who is capable of and willing to assume responsibility for facilitating subject compliance with study procedures
* All females of childbearing age and all sexually active males must agree to use an acceptable method of contraception throughout the study.

Exclusion Criteria:

* Use of any investigational drug within 30 days
* Use of prohibited medications
* Uncontrolled infection
* Active GI bleeding or a history of GI bleeding requiring blood transfusion (> 2 units) within 3 months
* Transjugular intrahepatic portosystemic shunt (TIPS) placement or revision within the past 90 days
* Recreational drug use or alcohol consumption for subjects with a history of alcohol or drug abuse within 6 months
* Lactating and/or pregnant females
* Active malignancy
* Clinically significant bowel disease, including obstruction, inflammatory bowel disease, or malabsorption
* Expected to undergo transplantation within 6 months
* Model for end-stage liver disease (MELD) score of > 25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (28):
- United States (28):
  - Stanford University Medical Center, Division of Gastroenterology and Hepatology, Palo Alto, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami / Center for Liver Diseases, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Health Science Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Hospital / Department of Gastroenterology, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Concorde Medical Group PLLC, New York, New York
  - NYU Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center / Center for Liver Disease and Transplantation, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - New York Medical College / Westchester Medical Center, Valhalla, New York
  - University of Cincinnati / Division of Digestive Diseases, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Digestive Disease Center at Vanderbilt, Nashville, Tennessee
  - Methodist Dallas Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine-St. Luke's Episcopal Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Result] Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Alexeeva O, Zupanets IA, Grinevich V, Baranovsky A, Dudar L, Fadieienko G, Kharchenko N, Klaryts'ka I, Morozov V, Grewal P, McCashland T, Reddy KG, Reddy KR, Syplyviy V, Bass NM, Dickinson K, Norris C, Coakley D, Mokhtarani M, Scharschmidt BF; HALT-HE Study Group. Randomized, double-blind, controlled study of glycerol phenylbutyrate in hepatic encephalopathy. Hepatology. 2014 Mar;59(3):1073-83. doi: 10.1002/hep.26611. PMID 23847109
- [Derived] Mokhtarani M, Diaz GA, Rhead W, Berry SA, Lichter-Konecki U, Feigenbaum A, Schulze A, Longo N, Bartley J, Berquist W, Gallagher R, Smith W, McCandless SE, Harding C, Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Dickinson K, Moors T, Norris C, Coakley D, Milikien DA, Nagamani SC, Lemons C, Lee B, Scharschmidt BF. Elevated phenylacetic acid levels do not correlate with adverse events in patients with urea cycle disorders or hepatic encephalopathy and can be predicted based on the plasma PAA to PAGN ratio. Mol Genet Metab. 2013 Dec;110(4):446-53. doi: 10.1016/j.ymgme.2013.09.017. Epub 2013 Oct 8. PMID 24144944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A enrollment: 01 December 2009 to 24 February 2010 Part B enrollment: 01 June 2010 to 31 October 2011
Pre-assignment Details: The study consisted of Part A, an open-label, dose-escalation lead-in to assess HPN-100 safety and PK, followed by Part B, a randomized, placebo controlled study to assess safety and efficacy of HPN-100.
Groups:
- HPN-100 6 mL and 9 mL: Subjects will undergo a one step dose escalation over 4 weeks. Subjects will initially receive 6 mL HPN-100 BID for 1 week. On Day 7 and following a satisfactory safety assessment of the subject, the dose will be escalated to 9 mL BID for an additional 3 weeks.
- HPN-100 6 mL: Subjects will receive 6 mL BID HPN-100 for 16 weeks (Part B)
- Placebo: Subjects will receive 6 mL BID placebo for 16 weeks (Part B)
Period: Part A: Open Label Safety run-in
Arm/Group | HPN-100 6 mL and 9 mL | HPN-100 6 mL | Placebo
Started | 15 | 0 | 0
Received 9 mL BID | 15 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Met protocol defined stopping rule | 4 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Period: Part B: Randomized, Placebo Controlled
Arm/Group | HPN-100 6 mL and 9 mL | HPN-100 6 mL | Placebo
Started | 0 | 90 (4 subjects who participated in Part A enrolled in Part B and remainder were newly enrolled) | 88
Completed | 0 | 55 | 67
Not Completed | 0 | 35 | 21
Not completed — Met protocol defined stopping rule | 0 | 19 | 16
Not completed — Withdrawal by Subject | 0 | 7 | 4
Not completed — Adverse Event | 0 | 6 | 1
Not completed — Noncompliance | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Physician stopped drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only the baseline characteristics of the subjects enrolled in Part B are presented.
Groups:
- HPN-100; Placebo: 6 mL BID
- Total: Total of all reporting groups
Arm/Group | HPN-100 | Placebo | Total
Number analyzed (Participants) | 90 | 88 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 78 | 163
  >=65 years | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (8.94) | 55.4 (8.85) | 54.6 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 29 | 74
  Male | 45 | 59 | 104
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88
  Russian Federation | 26 | 24 | 50
  Ukraine | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part A: The Rate of AEs and Tolerability of HPN-100
Description: Part A: The rate of AEs and tolerability of 6 mL and 9 mL doses of HPN-100 were considered the primary safety endpoints for Part A. Safety assessments included adverse events, laboratory tests (including ammonia, hematology, coagulation, liver function and serum chemistry parameters), vital signs, physical and neurological examinations, and electrocardiograms.
Time Frame: Part A: 28 days
Population: Safety population
Measure: Number; unit: Subjects
Groups:
- HPN-100 BID: 6 mL or 9 mL BID HPN-100 (Part A)
Arm/Group | HPN-100 BID
Number analyzed (Participants) | 15
Subjects
  Any AE | 11
  Gastrointestinal disorders | 9
  Metabolism and nutrition disorders | 7
  Infection and infestations | 4
  Nervous system disorders | 4
  Blood and lymphatic system disorders | 2
  Injury, poisoning and procedural complications | 2
  Musculoskeletal and connective tissue disorders | 2
  Psychiatric disorders | 2
  Any SAE | 5
  Death | 2

2. Secondary Outcome: Total Number of HE Events
Description: Secondary efficacy endpoint. The total number of HE events during the treatment phase for subjects in the placebo and active arms.
Time Frame: 112 Days
Population: Intent to treat (ITT)
Measure: Number; unit: HE event
Arm/Group | HPN-100 | Placebo
Number analyzed (Participants) | 90 | 88
HE event | 35 | 57
Statistical Analysis 1: Comparison: HPN-100 vs Placebo; Test type: Superiority or Other; p = 0.0354, Poisson regression adjusting for country

3. Primary Outcome: Part B: Proportion of Subjects Who Exhibit an HE Episode, Defined as Either of the Following During the Treatment Phase: WH ≥2; WH Grade and Asterixis Grade Increase of 1 Each, if Baseline WH = 0
Description: An HE event was defined as occurrences of either a West Haven (WH) Grade ≥2 or a WH Grade 1 and asterixis grade increase of 1 (if baseline WH = 0).
  The WH criteria are widely used for rating the severity of HE and are summarized below:
  Grade 1: trivial lack of awareness, euphoria or anxiety, shortened attention span, impaired performance of addition Grade 2: lethargy or apathy, minimal disorientation for time or place, subtle personality change, inappropriate behavior, impaired performance of subtraction Grade 3: somnolence to semi-stupor but responsive to verbal stimuli, confusion, gross disorientation Grade 4: coma (unresponsive to verbal or noxious stimuli)
  Asterixis was assessed after arm and forearm extension along with wrist dorsiflexion for 30 seconds and assigned a grade according to the following criteria:
  Grade 1: rare flaps Grade 2: occasional irregular flaps Grade 3: frequent flaps Grade 4: continuous flaps
Time Frame: Part B: 112 Days
Population: Intent to Treat (ITT)
Measure: Number; unit: participants
Groups:
- HPN-100: HPN-100 6 mL BID (Part B)
- Placebo: Placebo 6 mL BID (Part B)
Arm/Group | HPN-100 | Placebo
Number analyzed (Participants) | 90 | 88
participants | 19 | 32
Statistical Analysis 1: Comparison: HPN-100 vs Placebo; Test type: Superiority or Other; p = 0.0214, Cochran-Mantel-Haenszel

4. Secondary Outcome: Time to Meeting the Primary Endpoint
Description: Secondary efficacy endpoint. The time to the first HE episode during the treatment period was calculated using the Kaplan-Meier method. Subjects who did not experience an HE episode were censored at the time of their last asterixis assessment. Subjects who had no post-randomization data for the primary endpoint were considered to have an HE episode at Day 1.
Time Frame: 112 Days
Population: Intent to treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | HPN-100 | Placebo
Number analyzed (Participants) | 90 | 88
Days | NA [NA to NA] — Data are based on Kaplan-Meier point estimates. Because of low event rate (21.1%) it is not possible to estimate the median. | NA [NA to NA] — Data are based on Kaplan-Meier point estimates. Because of low event rate (36.4%) it is not possible to estimate the median
Statistical Analysis 1: Comparison: HPN-100 vs Placebo; Test type: Superiority or Other; p = 0.047, Regression, Cox; Hazard Ratio (HR) = 0.56

5. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Score
Description: Changes from Baseline to Day 56 and the Final Visit were compared between treatment groups using an ANCOVA model for the total index RBANS score ). The index score is a sum of the scores for each of the 5 individual domains (immediate memory, visuospatial/constructional, language, attention). The minimum and maximum total index scores are 40 and 160, respectively; a higher score is better.
Time Frame: Day 56, Final Visit (D112)
Population: Intent to treat (ITT)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HPN-100 | Placebo
Number analyzed (Participants) | 90 | 88
units on a scale
  Change from Baseline to D56 (Total Score) | -0.5 (1.54) | 3.2 (1.37)
  Change from Baseline to Final Visit (Total Score) | -10.7 (2.85) | -9.7 (3.33)
Statistical Analysis 1: Comparison: HPN-100 vs Placebo; Changes in the Total Index Score from Baseline and Day 56; Test type: Superiority or Other; p = 0.0713, ANCOVA
Statistical Analysis 2: Comparison: HPN-100 vs Placebo; Changes in the Total Index Score from Baseline and the Final Visit; Test type: Superiority or Other; p = 0.2520, ANCOVA

ADVERSE EVENTS:
Time Frame: Part A: 28 days Part B: 112 days
Groups:
- Part A: HPN-100: 6 mL BID for 7 days followed by 9 mL BID for 21 days, equivalent to approximately 13.2 and 19.8 grams of HPN-100/day, respectively
- Part B: HPN-100: 6 mL BID, equivalent to approximately 13.2 grams of HPN-100/day
- Part B: Placebo: Matching HPN-100 placebo, 6 mL BID
Arm/Group | Part A: HPN-100 | Part B: HPN-100 | Part B: Placebo
Serious Adverse Events (participants affected / at risk) | 5/15 | 20/90 | 12/88
Other Adverse Events (participants affected / at risk) | 11/15 | 71/90 | 67/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: HPN-100 (N=15) | Part B: HPN-100 (N=90) | Part B: Placebo (N=88)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Urinary tract infections (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: HPN-100 (N=15) | Part B: HPN-100 (N=90) | Part B: Placebo (N=88)
Nausea (Gastrointestinal disorders) | 2 (2) | 11 (11) | 13 (15)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 8 (8) | 9 (9)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (6)
Ascites (Gastrointestinal disorders) | 0 (0) | 5 (6) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 13 (14) | 7 (7)
Fatigue (Gastrointestinal disorders) | 0 (0) | 6 (6) | 7 (8)
Pyrexia (General disorders) | 0 (0) | 5 (5) | 3 (3)
AST increased (Investigations) | 0 (0) | 10 (11) | 5 (5)
ALT increased (Investigations) | 0 (0) | 8 (9) | 4 (4)
White blood cell count (WBC) decreased (Investigations) | 0 (0) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 8 (10) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other